CLINICAL TRIAL: NCT06296615
Title: Whether Vaginal Microbiota Affects Pregnancy Outcomes After Embryo Transfer
Status: Completed | Type: Observational
Sponsor: ShangHai Ji Ai Genetics & IVF Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-022
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Infertility, Female; Microbial Colonization
MeSH Terms: conditions — Infertility, Female; Communicable Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — vaginal secretion
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about vaginal microbial characteristics in the patients under in vitro fertilization treatment. The study aims to address the following questions: (1) Is there any difference in microbial composition between the pregnancy and non-pregnancy groups? (2) Is there any differences in specific bacterial species between the two groups? (3) What are the favorable or unfavorable profiles of vaginal microbiota associated with achieving pregnancy? Patients will be asked to complete a questionnaire regarding their basic characteristics, and vaginal secretions will be collected via vaginal swab during frozen-blastocyst transfer procedures. The study will compare vaginal microbiota between pregnant and non-pregnant patients to assess its potential influence on clinical outcomes.

DETAILED DESCRIPTION:
Despite clinicians' efforts to optimize clinical protocols in assisted reproduction, the clinical pregnancy rate continues to be unsatisfactory. Microbial dysbiosis has been implicated in numerous adverse reproductive conditions. The examination of microorganisms remains a promising avenue for improving clinical outcomes following embryo transfer in in-vitro fertilization (IVF) centers.

The vagina serves as the primary barrier, separating the external environment from the upper reproductive tract. Recent studies employing deep sequencing of microorganisms in IVF patients have shed light on the association between the diversity of vaginal microbiota and the abundance of specific microorganisms with crucial reproductive outcomes. However, certain studies have yielded inconsistent results, suggesting either no discernible association between vaginal microbiota and IVF outcomes or varying disparities in bacterial composition between groups with favorable and unfavorable clinical outcomes. Research into predictive models based on reproductive tract microbiota remains relatively limited. Hence, further studies are warranted to elucidate the correlation between vaginal microorganisms and pregnancy outcomes.

The aim of this study is to explore the characteristics of vaginal microbiota in patients undergoing IVF treatment and examine potential differences between those who achieve pregnancy and those who do not. Patients will be asked to complete a questionnaire regarding their basic characteristics, and vaginal secretions will be collected via vaginal swab during frozen-blastocyst transfer procedures. High-throughput sequencing of the V3-V4 variable region of the 16S rRNA gene will be conducted on the vaginal secretions of participants. Specifically, investigators will: (1) compare Alpha diversity between the two groups; (2) compare Beta diversity between the two groups; (3) investigate whether there are any differences in specific bacterial taxa between the two groups; (4) determine the favorable or unfavorable profiles of vaginal microbiota associated with achieving pregnancy; and (5) explore methods for predicting pregnancy outcomes based on vaginal microbiota. This study presents a prospective approach to utilizing microbial characteristics for predicting pregnancy outcomes before implementing further interventions, offering potential refinement of treatment strategies for IVF patients.

ELIGIBILITY:
Inclusion Criteria:

* Woman of 20-40 years of age
* Woman who have regular menstrual cycles and normal level of E2, P, FSH, LH, T, RPL in the early follicular phase
* Women who are scheduled for PGT cycles in IVF center and have a euploid blastocyst to transfer
* Women who have normal uterine and adnexal ultrasonography

Exclusion Criteria:

* embryos underwent double vitrification or a second biopsy
* patients having premature ovarian insufficiency (FSH > 12 mIU/ml and AMH < 1.1 ng/ml), abnormal uterine cavity, systemic disease, endometriosis American Fertility Score III/IV, or cancer
* those testing positive for mold spores or trichomonas in vaginal secretion examination and subjectively reported abnormal vaginal symptoms such as vaginal itching at 7 days before embryo transfer

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The patients who are under IVF treatment and have at least one high-quality euploid blastocysts to transfer. In addition, the participants should not have severe conditions that could adversely affect pregnancy outcomes, such as premature ovarian insufficiency or severe endometriosis.
Sampling Method: Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Rate of clinical pregnancy | 4 weeks after embryo transfer for the patient
  Clinical pregnancy is defined as the presence of a gestational sac confirmed by transvaginal ultrasound examination.

CONTACTS AND LOCATIONS:
Overall Officials: Yijuan Sun, Ph.D, Study Director — ShangHai Ji Ai Genetics & IVF Institute
Locations (1):
- Shanghai Ji Ai Genetics & IVF Institute, Shanghai, China

REFERENCES:
- [Result] Koedooder R, Singer M, Schoenmakers S, Savelkoul PHM, Morre SA, de Jonge JD, Poort L, Cuypers WJSS, Beckers NGM, Broekmans FJM, Cohlen BJ, den Hartog JE, Fleischer K, Lambalk CB, Smeenk JMJS, Budding AE, Laven JSE. The vaginal microbiome as a predictor for outcome of in vitro fertilization with or without intracytoplasmic sperm injection: a prospective study. Hum Reprod. 2019 Jun 4;34(6):1042-1054. doi: 10.1093/humrep/dez065. PMID 31119299